CLINICAL TRIAL: NCT05100615
Title: Healing Assessment of Osseous Defects After Surgical Removal of Periapical Lesions in the Presence of Hydroxyapatite, Nanohydroxyapatite and Combination of Nanohydroxyapatite and Platelet-rich Fibrin. A Clinical Study
Brief Title: Healing Assessment of Osseous Defects After Surgical Removal of Periapical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Amira mohammed elkholly, phD student- Endodontic Departement, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 238
Record Dates: First submitted 2021-09-28; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Effects of the Elements
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hydroxyappatite (Other): hydroxyapatite powder used for enhancement of bone regeneration
  Interventions: Procedure: surgery
- nanohydroxyapatite (Other): nanohydroxyapatite powder used for enhancement of bone regeneration
  Interventions: Procedure: surgery
- PRF with nanohydroxyapatite (Other): platelet rich fibrin mixed with nanohydroxyapatite used for enhancement of bone regeneration
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — applying the graft inside bony defect after surgery

SUMMARY:
recruited patients with periapical lesions will be divided into three groups and surgically treated with three types of bone graft (hydroxyappatite, nanohydroxyappatite and PRF WITH NANOHYDROXTAPPATITE) and then evaluated for month, three months and six months for the healing of periapical bone

ELIGIBILITY:
Inclusion Criteria:

* The patient will be in range of 20-45 years of age at the time of treatment, having periapical lesions starting from 5mm or more in diameter related to failed endodontically treated single canaled teeth.

Exclusion Criteria:

* Any systemic debilitating disease such as:

Diabetes mellitus, renal disease, Liver disease or liver failure, Rheumatoid arthritis, Neoplastic disease or its treatment, chronic corticosteroid therapy, chronic hepatitis B or C , History of hepatitis A, pregnant females.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
healing of periapical lesion | interappointment at 1 month, 3 months and 6 months
  change in size of bony defect

CONTACTS AND LOCATIONS:
Locations (1):
- Amira mohammed fathy Elkholly, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes